CLINICAL TRIAL: NCT04952389
Title: Acupuncture Therapy for COVID-Related Olfactory Loss
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Janalee K. Stokken, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 21-003531
Record Dates: First submitted 2021-07-02; First posted 2021-07-07 (Actual); Results first posted 2024-03-12 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-02

CONDITIONS: Olfactory Dysfunction; COVID-19
MeSH Terms: conditions — COVID-19 | interventions — Acupuncture Therapy; Budesonide; Olfactory Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Acupuncture Therapy Group (Experimental): Subjects will undergo ten sessions of acupuncture therapy with a licensed acupuncturist in addition to the standard of care.
  Interventions: Device: Acupuncture Therapy; Drug: Budesonide; Other: Olfactory Training
- Standard of Care (Active Comparator): Subjects will be treated with two times daily budesonide rinses and olfactory (sense of smell) training. This is considered the current standard of care in the treatment of olfactory dysfunction.
  Interventions: Drug: Budesonide; Other: Olfactory Training

INTERVENTIONS:
Device: Acupuncture Therapy — Consists of two treatments per week for five weeks
  Arms: Acupuncture Therapy Group
Drug: Budesonide — Twice daily nasal rinses with steroid medication (budesonide)
Other: Olfactory Training — involves smelling 4 different essential oils (e.g. rose, lemon, clove, and eucalyptus) twice a day for 20 seconds each (after the nasal rinse)

SUMMARY:
This study is looking at the role of acupuncture as a treatment for olfactory dysfunction in patients who tested positive for COVID-19.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older.
* Patients with post-viral olfactory dysfunction > 4 weeks.
* History of positive COVID-19 PCR.

Exclusion Criteria:

* Less than 18 years of age.
* Active sinus infection.
* New diagnosis of untreated CRS.
* Prior diagnosis of dementia or Parkinson's disease.
* Prior head trauma or neurosurgical procedure resulting in olfactory loss.
* Patients who do not speak or read English.
* Patients unable to understand and sign the study consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2021-12-07 (Actual); Primary Completion 2023-04-21 (Actual); Study Completion 2023-06-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janalee Stokken, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials

RESULTS

PARTICIPANT FLOW:
Groups:
- Acupuncture Therapy Group: Subjects underwent ten sessions of acupuncture therapy with a licensed acupuncturist in addition to the standard of care.
  Acupuncture Therapy: Consisted of two treatments per week for five weeks
  Budesonide: Twice daily nasal rinses with steroid medication (budesonide)
  Olfactory Training: involved smelling 4 different essential oils (e.g. rose, lemon, clove, and eucalyptus) twice a day for 20 seconds each (after the nasal rinse)
- Standard of Care: Subjects were treated with two times daily budesonide rinses and olfactory (sense of smell) training. This is considered the current standard of care in the treatment of olfactory dysfunction.
  Budesonide: Twice daily nasal rinses with steroid medication (budesonide)
  Olfactory Training: involved smelling 4 different essential oils (e.g. rose, lemon, clove, and eucalyptus) twice a day for 20 seconds each (after the nasal rinse)
Period: Overall Study
Arm/Group | Acupuncture Therapy Group | Standard of Care
Started | 15 | 15
Completed | 7 | 11
Not Completed | 8 | 4
Not completed — Withdrawal by Subject | 8 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Acupuncture Therapy Group | Standard of Care | Total
Number analyzed (Participants) | 15 | 15 | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 12 | 13 | 25
  >=65 years | 3 | 2 | 5
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 12 | 24
  Male | 3 | 3 | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 15 | 14 | 29
  Unknown or Not Reported | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 0 | 0 | 0
  White | 12 | 15 | 27
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 15 | 15 | 30

OUTCOME MEASURES:

1. Primary Outcome: Change in University of Pennsylvania Smell Identification Test (UPSIT) Scores
Description: The 40-item UPSIT is a measurement of the ability to detect odors where microencapsulated odorants on a strip are released by scratching. Each item is scored from 0 (did not correctly detect the odor) to 1 (correctly detected the odor). Total scores range from 0-40 with higher scores indicating better smell and lower scores indicating worse smell.
Time Frame: Baseline, post-treatment approximately 12 weeks
Population: Data not collected nor analyzed for eight subjects in the Acupuncture arm and four subjects in the Standard of Care arm
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Acupuncture Therapy Group | Standard of Care
Number analyzed (Participants) | 7 | 11
score on a scale | 2.571 (5.997) | 3.182 (5.306)

2. Secondary Outcome: Change in Patient-reported Subjective Olfactory Loss
Description: Patient-reported subjective olfactory loss measured by a 10-point visual analog scale with 10 representing no sense of smell and 1 representing normal smell.
Time Frame: Baseline, post-treatment approximately 12 weeks
Population: Data not collected nor analyzed for eight subjects in the Acupuncture arm and four subjects in the Standard of Care arm
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Acupuncture Therapy Group | Standard of Care
Number analyzed (Participants) | 7 | 11
score on a scale | 1.857 (2.167) | 1.727 (2.125)

3. Secondary Outcome: Change in Sino-Nasal Outcome Test (SNOT-22)
Description: Patient-reported subjective olfactory loss measured by SNOT-22 questionnaire, rating symptoms experiences from 0 = no problem, 5 = problem as bad as it can be, with a total score ranging of 0-110, lower scores indicate no problem and higher scores indicate more problem.
Time Frame: Baseline, post-treatment approximately 12 weeks
Population: Data not collected nor analyzed for eight subjects in the Acupuncture arm and four subjects in the Standard of Care arm
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Acupuncture Therapy Group | Standard of Care
Number analyzed (Participants) | 7 | 11
score on a scale | 7.143 (9.746) | 3.455 (15.035)

ADVERSE EVENTS:
Time Frame: Adverse Events were collected from baseline until end of study, approximately 3 months
Arm/Group | Acupuncture Therapy Group | Standard of Care
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/15
Other Adverse Events (participants affected / at risk) | 1/15 | 1/15
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Acupuncture Therapy Group (N=15) | Standard of Care (N=15)
Hyperglycemia (Metabolism and nutrition disorders) | 1 | 0
Brain fog (Nervous system disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-03-23): https://cdn.clinicaltrials.gov/large-docs/89/NCT04952389/Prot_SAP_000.pdf